CLINICAL TRIAL: NCT00777400
Title: A Pilot Trial to Assess the Effect of CNI Conversion to Efalizumab in T Regulatory Cells in Renal Transplantation
Brief Title: Pilot Trial to Assess Effect of CNI Conversion of Efalizumab on T Reg Cells
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: New safety information reported in the post-marketing setting with efalizumab for treatment of chronic plaque psoriasis and trial conduct feasibility issues.
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ACD4520 Efalizumab; ACD4520
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Autoimmune Diseases
Keywords: Kidney transplant; T regulatory cells; Efalizumab; Rejection; Safely convert renal transplant from mycophenolate mofetil and Calcineurin inhibitor to efalizumab and sirolimus
MeSH Terms: conditions — Autoimmune Diseases; Rejection, Psychology | interventions — efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Efalizumab will be started on Day 0 until the end of the study at Week 24. At the end of the first week, after efalizumab is started, cyclosporine or tacrolimus will be decreased by 50% and at 2 weeks the dose of cyclosporine or tacrolimus will be completely discontinued. At 12 weeks Cellcept or myfortic will be discontinued and the patient will be converted to sirolimus for the remainder of the study.
  Interventions: Drug: Efalizumab

INTERVENTIONS:
Drug: Efalizumab — 1 mg/kg of efalizumab administered sub q once weekly

SUMMARY:
The purpose of this pilot trial is to determine whether a conversion from calcineurin inhibitors (CNI) and mycophenolate mofetil (MMF) to a regimen consisting of efalizumab and sirolimus is associated with an increase in T regulatory cells, white cells that control the immune system and can prevent autoimmune diseases like arthritis or rejection of foreign organs,and does not result in an increase in acute rejection.

DETAILED DESCRIPTION:
The objective of this pilot trial is to determine whether the conversion from calcineurin inhibitors (CNI) and mycophenolate mofetil (MMF) to efalizumab and sirolimus is associated with an increase in T regulatory cells and does not result in an increase in acute rejection following conversion. CNIs are associated with progressive nephrotoxicity, increased cardiovascular risk factor as well as an inhibitory effect on T regulatory cells.

PRIMARY OBJECTIVE:

To determine if the combination of efalizumab and sirolimus results in a significant increase in T regulatory cells. A hundred percent increase in T regulatory cells will be determined to be an important biologic effect of the combination of efalizumab and sirolimus.

SECONDARY OBJECTIVES:

To assess the feasibility of the conversion from CNI/MMF to efalizumab/sirolimus and to determine that this combination is safe and effective

To determine if there is an increase in FoxP3 mRNA in the urine of converted patients. Urine FoxP3 is believed to correlate with T regs in the kidney.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Male or female, 18-70 years
* Recipients of primary renal transplants from living and deceased donors
* Stable renal function for 4 weeks prior to entry into the study
* No history of acute rejection
* Pretransplant negative crossmatch
* Hematocrit >30% at the time of inclusion, platelet count >100,000 and WBC ≥ 3.0
* If a female of childbearing potential, a negative pregnancy test and commitment to the use of two forms of effective contraception (birth control) for the duration of the study are necessary.
* If a non-sterile male, commitment to the use of two forms of effective contraception (birth control) for the duration of the study is necessary.

Exclusion Criteria:

* Patients with known hypersensitivity to Raptiva® (efalizumab) or any of its components.
* Pregnant or lactating women
* Pretransplant PRA >20%
* cGFR < 35/ml/min
* >500 mg protein as estimated by spot protein/creatinine ratio
* Recipients of other organ transplants
* Subject has a current malignancy or a history of malignancy, except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* Patients receiving experimental immunosuppressive agents
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Participation in another simultaneous medical investigation or trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine if the combination of efalizumab and sirolimus results in a significant increase in T regulatory cells. | Month 6

SECONDARY OUTCOMES:
The successful conversion from CNI to non-CNI regimen without increasing the rejection rate by more than 20%. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Nankivell BJ, Borrows RJ, Fung CL, O'Connell PJ, Allen RD, Chapman JR. The natural history of chronic allograft nephropathy. N Engl J Med. 2003 Dec 11;349(24):2326-33. doi: 10.1056/NEJMoa020009. PMID 14668458
- [Result] Meier-Kriesche HU, Schold JD, Srinivas TR, Kaplan B. Lack of improvement in renal allograft survival despite a marked decrease in acute rejection rates over the most recent era. Am J Transplant. 2004 Mar;4(3):378-83. doi: 10.1111/j.1600-6143.2004.00332.x. PMID 14961990
- [Result] Vincenti F, Mendez R, Pescovitz M, Rajagopalan PR, Wilkinson AH, Butt K, Laskow D, Slakey DP, Lorber MI, Garg JP, Garovoy M. A phase I/II randomized open-label multicenter trial of efalizumab, a humanized anti-CD11a, anti-LFA-1 in renal transplantation. Am J Transplant. 2007 Jul;7(7):1770-7. doi: 10.1111/j.1600-6143.2007.01845.x. PMID 17564637